CLINICAL TRIAL: NCT02306460
Title: Frontal Cognitive Control Functions Before and After Percutaneous Catheter Procedures in Treatment of Atrial Fibrillation
Status: Terminated | Type: Observational
Why Stopped: Changes in personnel
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kati Järvelä, MD, PhD, Tampere University Hospital
Other Study IDs: R14068
Record Dates: First submitted 2014-07-11; First posted 2014-12-03 (Estimated); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Neurobehavioral Manifestations; Atrial Fibrillation
Keywords: Neurobehavioral Manifestations; POCD; Atrial Fibrillation; Anti-Arrhythmia; Atrial Appendage Closure
MeSH Terms: conditions — Neurobehavioral Manifestations; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- left atrial catheter ablation
- left atrial appendix closure
- paroxysmal atrial fibrillation control group
- persistent atrial fibrillation control group

SUMMARY:
Atrial fibrillation is a common arrythmia. It is an independent risk factor for stroke. There for anticoagulation therapy is used for atrial fibrillation patients. Alternatively, left atrial appendix closure can be used, if the risk for bleeding complications is deemed greater than the possible antithrombotic benefit of anticoagulation medication. Up to 70% of ischemic complications can be prevented with anticoagulation therapy, and left atrial appendix closure seems to have comparable results. Also left atrial catherter ablation (LACA) is gaining popularity as a therapeutic intervention for atrial fibrillation.

However, the procedure is associated with 0,5-1% perioperative risk of clinically evident transient ischemic attack (TIA) or stroke. While the incidence of clinically evident ischemic complications remain relatively low, recent data suggest that 13%-20% of patients undergoing LACA are affected by post-operative neurocognitive dysfunction (POCD) 90 days after ablation.

The goal of the study is to improve detection of subtle brain dysfunction after cardiac interventions by employing an experimental executive reaction time (RT) test along with EEG recording in aims to improve objective detection of subtle brain dysfunction assumed to underlie persistent cognitive, somatic, and affective complaints reported by patients who have undergone atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

* age 50-70
* undergoing left atrial catheter ablation or percutaneous left atrial appendix closure procedure
* In the ablation group, patients will qualify for the study if they have symptomatic atrial fibrillation (EHRA classification 2-4) and if their risk of thromboembolic complications with CHA2DS2VASc scale is low (0-2 points).

Exclusion Criteria:

* Age under 18 or over 70 years.
* Contraindication for anticoagulation therapy (in ablation group),
* Previous neurological or psychiatric disorder.
* Significant visual problem that can't be corrected for,
* problems with upper arm/hand use, that would make the execution of the test difficult.
* normal contraindications for the ablation and appendix closure procedures.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 80 patients will be drafted for the study. The subjects will be recruited from Tampere University Hospital Heart Hospital Co. Total of fifty patients, men and women between 50-70 years, undergoing left atrial catheter ablation (LACA) (30 patients) or percutaneous left atrial appendix closure procedure (20 patients) because of paroxysmal or persistent atrial fibrillation, will be recruited for the study.
  A control group of 15 patients with paroxysmal atrial fibrillation and 15 patients with persistent atrial fibrillation who are treated with antiarrhythmic and anticoagulation therapies suggested by current guidelines will be tested with the same testing schema and time points. Control group will be drafted from the cardiologic patients of the Heart Hospital and also from Hatanpää Hospital cardiologic outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-02-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Changes in response speeds (ms) and response error rate (%) in the executive RT-test | 1 day before procedure, 3 months and 1 year after post-procedure

SECONDARY OUTCOMES:
Changes in amplitude of N2/P3 complex in the EEG recording | 1 day before procedure, 3 months and 1 year after post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa Hartikainen, MD, Docent, Study Director — Behavioral Neurology Research Unit; Kati Järvelä, MD, PhD, Study Director — Tampere Heart Hospital; Arvi Yli-Hankala, MD, Professor, Study Director — Tampere University Hospital; Jonne Liimatainen, MD, Principal Investigator — Tampere University Hospital; Pekka Raatikainen, MD, Docent, Study Director — Tampere Heart Hospital; Jaakko Inkovaara, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Heart Hospital, Tampere, Finland